CLINICAL TRIAL: NCT00115791
Title: A Phase 3, Prospective, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Tolerance and Efficacy Study of RSD1235 in Subjects With Atrial Fibrillation or Atrial Flutter
Brief Title: Study to Determine the Response and Effectiveness of RSD1235 in Subjects With Atrial Fibrillation or Atrial Flutter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Advanz Pharma (Industry)
Responsible Party: Sr Manager Clinical Trial Registry, Astellas Pharma US, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-7-010; Cardiome 1235-0504
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Atrial Flutter; Atrial Fibrillation
Keywords: Atrial Flutters; Atrial Fibrillations; RSD1235
MeSH Terms: conditions — Atrial Flutter; Atrial Fibrillation | interventions — vernakalant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RSD1235
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RSD1235 — IV
  Other Names: vernakalant; Kynapid
  Arms: 1
Drug: placebo — IV
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of RSD1235 compared with placebo, in the conversion of atrial fibrillation or atrial flutter to sinus rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Atrial flutter or atrial fibrillation that has been sustained for greater than 3 hours and up to 45 days

Exclusion Criteria:

* Myocardial infarction, acute coronary syndrome or cardiac surgery within 30 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of RSD1235 compared with placebo, in the conversion of atrial fibrillation or atrial flutter to sinus rhythm | Infusion plus 1.5 hours

SECONDARY OUTCOMES:
To assess the time taken from exposure to first treatment to first conversion to sinus rhythm | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (48):
- United States (19):
  - Investigative Site, Birmingham, Alabama
  - Investigative Site, Huntsville, Alabama
  - Investigative Site, Gainesville, Florida
  - Investigative Site, Orlando, Florida
  - Investigative Site, Port Charlotte, Florida
  - Investigative Site, Indianapolis, Indiana
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Lansing, Michigan
  - Investigative Site, Petoskey, Michigan
  - Investigative Site, Saint Paul, Minnesota
  - Investigative Site, Tupelo, Mississippi
  - Investigative Site, Holmdel, New Jersey
  - Investigative Site, Cincinnati, Ohio
  - Investigative Site, Amarillo, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Richmond, Virginia
  - Investigative Site, Tacoma, Washington
  - Investigative Site, Marshfield, Wisconsin
- Argentina (2):
  - Investigative Site, Buenos Aires
  - Investigative Site, Mendoza
- Canada (7):
  - Investigative Site, Calgary, Alberta
  - Investigative Site, Edmonton, Alberta
  - Investigative Site, Halifax, Nova Scotia
  - Investigative Site, Ottawa, Ontario
  - Investigative Site, Toronto, Ontario
  - Investigative Site, Montreal, Quebec
  - Investigative Site, Terrebonne, Quebec
- Investigative Site, Santiago, Cironaria, Chile
- Denmark (13):
  - Investigative Site, Aalborg
  - Investigative Site, Arhus C
  - Investigative Site, Esbjerg
  - Investigative Site, Fredericia
  - Investigative Site, Frederikssund
  - Investigative Site, Herlev
  - Investigative Site, Hjørring
  - Investigative Site, Holstebro
  - Investigative Site, Horsens
  - Investigative Site, Hvidovre
  - Investigative Site, København NV
  - Investigative Site, København S
  - Investigative Site, Køge
- Investigative Site, Magdalena de las Salinas, Mexico
- Sweden (5):
  - Investigative Site, Malmo
  - Investigative Site, Mölndal
  - Investigative Site, Örebro
  - Investigative Site, Stockholm
  - Investigative Site, Uppsala